CLINICAL TRIAL: NCT00051363
Title: APPLES: Apnea Positive Pressure Long-Term Efficacy Study
Brief Title: Apnea Positive Pressure Long-Term Efficacy Study
Acronym: APPLES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Clete A. Kushida, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150; U01HL068060 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-13 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes; Sleep
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active CPAP (Active Comparator): Active Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: Active CPAP
- Sham CPAP (Placebo Comparator): Sham Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: Sham CPAP

INTERVENTIONS:
Device: Active CPAP — Nightly nasal continuous positive airway pressure (CPAP)
  Other Names: Positive Pressure Respiration
  Arms: Active CPAP
Device: Sham CPAP — Sham CPAP machine will be used for participants in the placebo group.
  Other Names: Sham CPAP machine
  Arms: Sham CPAP

SUMMARY:
The purpose of this study is to determine the effectiveness of nasal continuous positive airway pressure (CPAP) therapy for the treatment of obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
BACKGROUND:

Nasal CPAP therapy is in widespread use as the primary treatment for OSAS, a sleep-related breathing disorder affecting more than 15 million Americans. The therapeutic effectiveness of CPAP in providing significant, stable, and long-term neurocognitive or other functional benefits to patients with OSAS has not been systematically investigated.

DESIGN NARRATIVE:

The study is a randomized, blinded, sham-controlled, multi-center trial of CPAP therapy. The principal aims of the study are: 1) to assess the long-term effectiveness of CPAP therapy on neurocognitive function, mood, sleepiness, and quality of life by administering tests of these indices to subjects randomly assigned to active or sham CPAP; 2) to identify specific neurocognitive deficits associated with OSAS in a large, heterogeneous subject population; 3) to determine which deficits in neurocognitive function in OSAS subjects are reversible and most sensitive to the effects of CPAP; 4) to develop a composite multivariate outcome measure from the results of this study that can be used to assess the clinical effectiveness of CPAP in improving neurocognitive function, mood, sleepiness, and quality of life; and 5) to use functional magnetic resonance imaging to compare cortical activation before and after CPAP therapy, and to assess whether this change is associated with improvement in specific neurocognitive task performance. The primary endpoint of the study is the effect of six months of CPAP treatment on neurocognitive function. A total of 1100 subjects (550 per treatment group) will be enrolled from the patient populations at five sites (Stanford University; University of Arizona; Brigham and Women's Hospital; Massachusetts; St. Luke's Hospital, Missouri; St. Mary Medical Center, Washington).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults age 18 years or older with a diagnosis of OSAS using clinical criteria defined by the study protocol
* Study participation may require seven or more laboratory visits over six months

Exclusion Criteria:

* Prior treatment for OSAS with continuous positive airway pressure or surgery
* Potential sleep apnea complications that may affect the health or safety of the participant, including low blood oxygen, recent near-miss or prior automobile accident due to sleepiness, congestive heart failure, history of angina, coronary artery disease, myocardial infarction or stroke, cardiac rhythm disturbance, and chronic neurological disorders affecting neurocognitive abilities or daily function
* The use of hypnotics, anxiolytics, sedating antidepressants, anticonvulsants, sedating antihistamines, stimulants or other medications likely to affect neurocognitive function and/or alertness
* Respiratory disease requiring medications (unless on stable medications for 2 months)
* Cancer, unless in remission for greater than one year and not taking exclusionary medications
* Self-reported renal failure
* Pregnancy anytime during a subject's participation
* Psychiatric illness, as defined by a DSM-IV diagnosis, except for depression or mild anxiety
* Narcolepsy, idiopathic hypersomnolence, DSM-IV chronic insomnia, restless legs syndrome, or rapid eye movement (REM) behavior disorder
* Current use of diurnal or nocturnal supplemental oxygen
* Significant vision, hearing, or coordination problems
* Difficulty understanding or speaking English
* Currently working night or rotating shifts
* Consumption of more than 10 caffeinated beverages per day (approximately 1,000 mg per day)
* Smokers whose habit interferes with the overnight polysomnogram or with the battery of testing during the day
* Consumption of more than 2 alcoholic beverages per day
* Any illicit drug usage or marijuana usage more than once a week
* Any individual in the household currently on CPAP or on CPAP in the past
* A score of 26 or less on the Mini Mental State Examination (MMSE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2002-09; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Dement, MD, PhD, Study Chair — Stanford University; Clete A. Kushida, MD, PhD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - University of Arizona AHSC, Tucson, Arizona
  - Stanford University School of Medicine, Palo Alto, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - St. Luke's Hospital, Chesterfield, Missouri
  - St. Mary Medical Center, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: Yes
Only in de-identified format to researchers

REFERENCES:
- [Background] Kushida CA, Nichols DA, Quan SF, Goodwin JL, White DP, Gottlieb DJ, Walsh JK, Schweitzer PK, Guilleminault C, Simon RD, Leary EB, Hyde PR, Holmes TH, Bloch DA, Green S, McEvoy LK, Gevins A, Dement WC. The Apnea Positive Pressure Long-term Efficacy Study (APPLES): rationale, design, methods, and procedures. J Clin Sleep Med. 2006 Jul 15;2(3):288-300. PMID 17561541
- [Background] Holmes TH, Nichols DA, Thomander D, Kushida CA. A method for estimating normative distributions for study-specific populations of clinical trials. Contemp Clin Trials. 2012 Mar;33(2):445-9. doi: 10.1016/j.cct.2011.11.014. Epub 2011 Nov 25. PMID 22138103
- [Background] Gevins A, Smith ME, McEvoy LK, Ilan AB, Chan CS, Jiang A, Sam-Vargas L, Abraham G. A cognitive and neurophysiological test of change from an individual's baseline. Clin Neurophysiol. 2011 Jan;122(1):114-20. doi: 10.1016/j.clinph.2010.06.010. Epub 2010 Jul 8. PMID 20619727
- [Result] Quan SF, Chan CS, Dement WC, Gevins A, Goodwin JL, Gottlieb DJ, Green S, Guilleminault C, Hirshkowitz M, Hyde PR, Kay GG, Leary EB, Nichols DA, Schweitzer PK, Simon RD, Walsh JK, Kushida CA. The association between obstructive sleep apnea and neurocognitive performance--the Apnea Positive Pressure Long-term Efficacy Study (APPLES). Sleep. 2011 Mar 1;34(3):303-314B. doi: 10.1093/sleep/34.3.303. PMID 21358847
- [Result] Kushida CA, Nichols DA, Holmes TH, Quan SF, Walsh JK, Gottlieb DJ, Simon RD Jr, Guilleminault C, White DP, Goodwin JL, Schweitzer PK, Leary EB, Hyde PR, Hirshkowitz M, Green S, McEvoy LK, Chan C, Gevins A, Kay GG, Bloch DA, Crabtree T, Dement WC. Effects of continuous positive airway pressure on neurocognitive function in obstructive sleep apnea patients: The Apnea Positive Pressure Long-term Efficacy Study (APPLES). Sleep. 2012 Dec 1;35(12):1593-602. doi: 10.5665/sleep.2226. PMID 23204602
- [Result] Vasquez MM, Goodwin JL, Drescher AA, Smith TW, Quan SF. Associations of dietary intake and physical activity with sleep disordered breathing in the Apnea Positive Pressure Long-Term Efficacy Study (APPLES). J Clin Sleep Med. 2008 Oct 15;4(5):411-8. PMID 18853696
- [Result] Quan SF, Budhiraja R, Clarke DP, Goodwin JL, Gottlieb DJ, Nichols DA, Simon RD, Smith TW, Walsh JK, Kushida CA. Impact of treatment with continuous positive airway pressure (CPAP) on weight in obstructive sleep apnea. J Clin Sleep Med. 2013 Oct 15;9(10):989-93. doi: 10.5664/jcsm.3064. PMID 24127141
- [Result] Batool-Anwar S, Goodwin JL, Drescher AA, Baldwin CM, Simon RD, Smith TW, Quan SF. Impact of CPAP on activity patterns and diet in patients with obstructive sleep apnea (OSA). J Clin Sleep Med. 2014 May 15;10(5):465-72. doi: 10.5664/jcsm.3686. PMID 24910546
- [Result] Quan SF, Budhiraja R, Batool-Anwar S, Gottlieb DJ, Eichling P, Patel S, Shen W, Walsh JK, Kushida CA. Lack of Impact of Mild Obstructive Sleep Apnea on Sleepiness, Mood and Quality of Life. Southwest J Pulm Crit Care. 2014;9(1):44-56. doi: 10.13175/swjpcc082-14. PMID 25232509
- [Result] Quan SF, Budhiraja R, Clarke DP, Goodwin JL, Gottlieb DJ, Nichols DA, Simon RD, Smith TW, Walsh JK, Kushida CA, Phillips B. You still need more than CPAP for OSA patients to lose weight. J Clin Sleep Med. 2014 Mar 15;10(3):349. doi: 10.5664/jcsm.3552. No abstract available. PMID 24634638
- [Result] Prilipko O, Huynh N, Thomason ME, Kushida CA, Guilleminault C. An fMRI study of cerebrovascular reactivity and perfusion in obstructive sleep apnea patients before and after CPAP treatment. Sleep Med. 2014 Aug;15(8):892-8. doi: 10.1016/j.sleep.2014.04.004. Epub 2014 May 4. PMID 24916094
- [Result] Huynh NT, Prilipko O, Kushida CA, Guilleminault C. Volumetric Brain Morphometry Changes in Patients with Obstructive Sleep Apnea Syndrome: Effects of CPAP Treatment and Literature Review. Front Neurol. 2014 Apr 29;5:58. doi: 10.3389/fneur.2014.00058. eCollection 2014. PMID 24808886
- [Result] Prilipko O, Huynh N, Schwartz S, Tantrakul V, Kushida C, Paiva T, Guilleminault C. The effects of CPAP treatment on task positive and default mode networks in obstructive sleep apnea patients: an fMRI study. PLoS One. 2012;7(12):e47433. doi: 10.1371/journal.pone.0047433. Epub 2012 Dec 5. PMID 23227139
- [Result] Prilipko O, Huynh N, Schwartz S, Tantrakul V, Kim JH, Peralta AR, Kushida C, Paiva T, Guilleminault C. Task positive and default mode networks during a parametric working memory task in obstructive sleep apnea patients and healthy controls. Sleep. 2011 Mar 1;34(3):293-301A. doi: 10.1093/sleep/34.3.293. PMID 21358846
- [Result] Budhiraja R, Kushida CA, Nichols DA, Walsh JK, Simon RD, Gottlieb DJ, Quan SF. Impact of Randomization, Clinic Visits, and Medical and Psychiatric Cormorbidities on Continuous Positive Airway Pressure Adherence in Obstructive Sleep Apnea. J Clin Sleep Med. 2016 Mar;12(3):333-41. doi: 10.5664/jcsm.5578. PMID 26518698
- [Result] Batool-Anwar S, Goodwin JL, Kushida CA, Walsh JA, Simon RD, Nichols DA, Quan SF. Impact of continuous positive airway pressure (CPAP) on quality of life in patients with obstructive sleep apnea (OSA). J Sleep Res. 2016 Dec;25(6):731-738. doi: 10.1111/jsr.12430. Epub 2016 May 30. PMID 27242272
- [Derived] Zinchuk AV, Kushida CA, Walker A, Wellman A, Azarbarzin A, Alex RM, Varga AW, Sands SA, Yaggi HK. Arousal threshold modifies the effect of CPAP on executive function among individuals with obstructive sleep apnoea. Eur Respir J. 2025 Feb 13;65(2):2401183. doi: 10.1183/13993003.01183-2024. Print 2025 Feb. PMID 39572221
- [Derived] Knauert MP, Adekolu O, Xu Z, Deng A, Chu JH, Baldassarri SR, Kushida C, Yaggi HK, Zinchuk A. Morning Chronotype Is Associated with Improved Adherence to Continuous Positive Airway Pressure among Individuals with Obstructive Sleep Apnea. Ann Am Thorac Soc. 2023 Aug;20(8):1182-1191. doi: 10.1513/AnnalsATS.202210-885OC. PMID 36917194
- [Derived] Batool-Anwar S, Omobomi O, Quan SF. The effect of CPAP on HRQOL as measured by the Quality of Well-Being Self Administered Questionaire (QWB-SA). Southwest J Pulm Crit Care. 2020;20(1):29-40. doi: 10.13175/swjpcc070-19. PMID 32190413
- [Derived] Holmes TH, Kushida CA. Adherence to continuous positive airway pressure improves attention/psychomotor function and sleepiness: a bias-reduction method with further assessment of APPLES. Sleep Med. 2017 Sep;37:130-134. doi: 10.1016/j.sleep.2017.06.022. Epub 2017 Jul 14. PMID 28899524

RESULTS

PARTICIPANT FLOW:
Groups:
- Active CPAP: Active Continuous Positive Airway Pressure (CPAP) is widely used for the treatment of Obstructive Sleep Apnea (OSA)
- Sham CPAP: Sham Continuous Positive Airway Pressure (CPAP) has been modified to be sub-therapeutic, yet closely simulates an Active CPAP device.
Period: Overall Study
Arm/Group | Active CPAP | Sham CPAP
Started | 558 | 547
Randomized & Analyzed | 556 | 542
Completed 2M Visit On-Treatment | 456 | 417
Completed 2M Visit On-Study | 468 | 432
Completed 6M Visit On-Treatment | 427 | 372
Completed 6M Vist On-Study | 443 | 403
Completed | 443 | 403
Not Completed | 115 | 144
Not completed — Dropped Post-Rand for Any Reason | 102 | 126
Not completed — Disqualified Post-Rand for Any Reason | 9 | 11
Not completed — Death | 2 | 2
Not completed — Excluded Pre-Randomization | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CPAP | Sham CPAP | Total
Number analyzed (Participants) | 556 | 542 | 1098
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 459 | 464 | 923
  >=65 years | 96 | 78 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (12.2) | 50.8 (12.2) | 51.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 186 | 379
  Male | 363 | 356 | 719
Region of Enrollment [Number; unit: participants]
  United States | 556 | 542 | 1098

OUTCOME MEASURES:

1. Primary Outcome: Effect of CPAP on Neurocognitive Function: E/F Function- SWMT-OMD
Description: There are three primary measures of neurocognitive function measured for APPLES, each representing a different domain: Executive and Frontal-lobe (E/F) Function- Sustained Working Memory Test Overall Mid-Day Index (SWMT-OMD), Attention and Psychomotor (A/P) Function- Pathfinder Number Test Total Time (PFN-TOTL), and Learning and Memory (L/M) Function- Buschke Selective Reminding Test Sum Recall (BSRT-SR).
  This is domain #1: Executive and Frontal-lobe (E/F) Function- Sustained Working Memory Test Overall Mid-Day Index (SWMT-OMD)
  SWMT-OMD is a scaled score that indicates whether the participant scored lower or higher relative to baseline using standard deviation units. It is computed as the mean of three sub-scores, one based on working memory (WM) task performance (behavioral WM sub-score: speed, accuracy), and the other two on electroencephalogram (EEG) (cortical activation sub-score: neural workload, attentional effort during WM task; alertness sub-score: resting alertness).
Time Frame: 2 months and 6 months post intervention
Population: Analyses conducted in accordance with the intention-to-treat principle.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
score on a scale
  SWMT-OMD 2M | 0.035 [-0.019 to 0.090] | -0.074 [-0.133 to -0.015]
  SWMT-OMD 6M | 0.072 [0.012 to 0.132] | 0.018 [-0.046 to 0.082]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M E/F Function- SWMT-OMD; Test type: Superiority or Other; p = 0.0074, Regression, Linear — 2M E/F Function- SWMT-OMD; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses). After correction for multiple comparisons (sequential Bonferroni) P Value=0.0444 (NS); Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M E/F Function- SWMT-OMD; Test type: Superiority or Other; p = 0.2254, Regression, Linear — 6M E/F Function- SWMT-OMD; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); Generalized Linear Models (GLM) were run by visit (2M and 6M)

2. Primary Outcome: Effect of CPAP on Neurocognitive Function: A/P Function- PFN-TOTL
Description: There are three primary measures of neurocognitive function measured for APPLES, each representing a different domain: Executive and Frontal-lobe (E/F) Function- Sustained Working Memory Test Overall Mid-Day Index (SWMT-OMD), Attention and Psychomotor (A/P) Function- Pathfinder Number Test Total Time (PFN-TOTL), and Learning and Memory (L/M) Function- Buschke Selective Reminding Test Sum Recall (BSRT-SR).
  This is domain #2: Attention and Psychomotor (A/P) Function- Pathfinder Number Test Total Time (PFN-TOTL)
Time Frame: Measured at diagnostic visit (baseline) and 2 months and 6 months post intervention
Population: Analyses conducted in accordance with the intention-to-treat principle.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
seconds
  PFN-TOTL Dx | 23.32 [22.88 to 23.78] | 23.08 [22.64 to 23.54]
  PFN-TOTL 2M | 23.56 [23.05 to 24.10] | 22.92 [22.41 to 23.45]
  PFN-TOTL 6M | 23.48 [22.98 to 24.00] | 23.01 [22.51 to 23.54]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX A/P Function- PFN-TOTL. Data were reciprocal transformed for analysis and back-transformed for reporting; Test type: Superiority or Other; p = 0.4538, Parametric survival analysis — DX A/P Function- PFN-TOTL; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); Parametric survival analyses were conducted using by-visit comparisons for A/P Function- PFN-TOTL since these data were right censored at 60
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M A/P Function- PFN-TOTL. Data were reciprocal transformed for analysis and back-transformed for reporting; Test type: Superiority or Other; p = 0.0860, Parametric survival analysis — 2M A/P Function- PFN-TOTL; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M A/P Function- PFN-TOTL. Data were reciprocal transformed for analysis and back-transformed for reporting; Test type: Superiority or Other; p = 0.2103, Parametric survival analysis — 6M A/P Function- PFN-TOTL; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); [statistical method as in outcome 2, analysis 1]

3. Primary Outcome: Effect of CPAP on Neurocognitive Function: L/M Function- BSRT-SR
Description: There are three primary measures of neurocognitive function measured for APPLES, each representing a different domain: Executive and Frontal-lobe (E/F) Function- Sustained Working Memory Test Overall Mid-Day Index (SWMT-OMD), Attention and Psychomotor (A/P) Function- Pathfinder Number Test Total Time (PFN-TOTL), and Learning and Memory (L/M) Function- Buschke Selective Reminding Test Sum Recall (BSRT-SR).
  This is domain #3: Learning and Memory (L/M) Function- Buschke Selective Reminding Test Sum Recall (BSRT-SR)
Time Frame: Measured at diagnostic visit (baseline) and 2 months and 6 months post intervention
Population: Analyses conducted in accordance with the intention-to-treat principle.
Measure: Mean (95% Confidence Interval); unit: number of words recalled
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
number of words recalled
  BSRT-SR Dx | 49.72 [48.95 to 50.48] | 49.86 [49.09 to 50.64]
  BSRT-SR 2M | 52.32 [51.50 to 53.13] | 51.95 [51.10 to 52.80]
  BSRT-SR 6M | 54.09 [53.26 to 54.91] | 54.28 [53.41 to 55.13]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX L/M Function- BSRT-SR; Test type: Superiority or Other; p = 0.7936, Regression, Linear — DX L/M Function- BSRT-SR; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M L/M Function- BSRT-SR; Test type: Superiority or Other; p = 0.5444, Regression, Linear — 2M L/M Function- BSRT-SR; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M L/M Function- BSRT-SR; Test type: Superiority or Other; p = 0.7569, Regression, Linear — 6M L/M Function- BSRT-SR; P<0.0307 indicates statistical significance for raw P values (after adjustment for O'Brien-Fleming spending across 3 interim analyses); Generalized Linear Models (GLM) were run by visit (2M and 6M)

4. Secondary Outcome: Attention and Psychomotor (A/P) Function: Pathfinder Number- Reaction Time (PN-RT)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Attention and Psychomotor (A/P) Function: Pathfinder Number- Reaction Time (PN-RT), Psychomotor Vigilance Task- Median Reaction Time (PVT-MedRT), and PVT- Mean Slowest 10% of Reaction Times (PVT-Slo10%RT).
  These data are for variable #1: Pathfinder Number- Reaction Time (PN-RT)
Time Frame: 2 months and 6 months post intervention
Population: Analyses conducted in accordance with the intention-to-treat principle. Analyses performed by OSA severity level categorized by apnea hypopnea index (AHI: # of respiratory events/hr of sleep) obtained via baseline polysomnography. Categories are: Mild OSA (AHI = 10-14.9; exclusion if AHI <10), Moderate OSA (AHI = 15-29.9), Severe OSA (AHI >=30).
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
seconds
  2M PN-RT Mild OSA | 0.811 [0.785 to 0.839] | 0.801 [0.774 to 0.830]
  2M PN-RT Moderate OSA | 0.831 [0.811 to 0.852] | 0.825 [0.806 to 0.845]
  2M PN-RT Severe OSA | 0.818 [0.802 to 0.834] | 0.812 [0.797 to 0.828]
  6M PN-RT Mild OSA | 0.811 [0.784 to 0.839] | 0.795 [0.767 to 0.826]
  6M PN-RT Moderate OSA | 0.830 [0.808 to 0.853] | 0.819 [0.799 to 0.841]
  6M PN-RT Severe OSA | 0.817 [0.800 to 0.836] | 0.806 [0.790 to 0.823]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M L/M Function- PN-RT. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ. A pre-randomization baseline PN-RT and months since randomization were also included as covariates; Test type: Superiority or Other; p = 0.5606, Mixed Models Analysis — 2M L/M Function- PN-RT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6487, Mixed Models Analysis — 2M L/M Function- PN-RT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5667, Mixed Models Analysis — 2M L/M Function- PN-RT (Severe OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 6M L/M Function- PN-RT. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ. A pre-randomization baseline PN-RT and months since randomization were also included as covariates; Test type: Superiority or Other; p = 0.3972, Mixed Models Analysis — 6M L/M Function- PN-RT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.3973, Mixed Models Analysis — 6M L/M Function- PN-RT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.3055, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 5]; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)

5. Secondary Outcome: Attention and Psychomotor (A/P) Function: Psychomotor Vigilance Task- Median Reaction Time (PVT-MedRT)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Attention and Psychomotor (A/P) Function: Pathfinder Number- Reaction Time (PN-RT), Psychomotor Vigilance Task- Median Reaction Time (PVT-MedRT), and PVT- Mean Slowest 10% of Reaction Times (PVT-Slo10%RT).
  These data are for variable #2: Psychomotor Vigilance Task- Median Reaction Time (PVT-MedRT)
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
milliseconds
  2M PVT-MedRT Mild OSA | 245.31 [230.94 to 260.58] | 253.89 [238.02 to 270.82]
  2M PVT-MedRT Moderate OSA | 248.68 [237.96 to 259.89] | 248.94 [237.99 to 260.40]
  2M PVT-MedRT Severe OSA | 243.25 [235.36 to 251.41] | 247.55 [238.79 to 256.62]
  6M PVT-MedRT Mild OSA | 245.23 [230.20 to 261.23] | 254.05 [237.26 to 272.03]
  6M PVT-MedRT Moderate OSA | 248.60 [236.74 to 261.04] | 249.10 [236.95 to 261.86]
  6M PVT-MedRT Severe OSA | 243.17 [234.05 to 252.64] | 247.70 [237.46 to 258.38]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M A/P Function- PVT-MedRT. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ. Months since randomization were also included as covariate; Test type: Superiority or Other; p = 0.3699, Mixed Models Analysis — 2M A/P Function- PVT-MedRT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9673, Mixed Models Analysis — 2M A/P Function- PVT-MedRT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3426, Mixed Models Analysis — 2M A/P Function- PVT-MedRT (Severe OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3901, Mixed Models Analysis — 6M A/P Function- PVT-MedRT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9464, Mixed Models Analysis — 6M A/P Function- PVT-MedRT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4372, Mixed Models Analysis — 6M A/P Function- PVT-MedRT (Severe OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)

6. Secondary Outcome: Attention and Psychomotor (A/P) Function: PVT- Mean Slowest 10% of Reaction Times (PVT-Slo10%RT)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Attention and Psychomotor (A/P) Function: Pathfinder Number- Reaction Time (PN-RT), Psychomotor Vigilance Task- Median Reaction Time (PVT-MedRT), and PVT- Mean Slowest 10% of Reaction Times (PVT-Slo10%RT).
  These data are for variable #3: PVT- Mean Slowest 10% of Reaction Times (PVT-Slo10%RT)
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
milliseconds
  2M PVT-Slo10%RT Mild OSA | 403.00 [375.99 to 431.95] | 402.32 [376.77 to 429.62]
  2M PVT-Slo10%RT Moderate OSA | 412.44 [390.91 to 435.16] | 407.84 [387.67 to 429.06]
  2M PVT-Slo10%RT Severe OSA | 400.57 [384.51 to 417.30] | 406.11 [387.05 to 426.07]
  6M PVT-Slo10%RT Mild OSA | 396.87 [370.79 to 424.79] | 401.28 [375.51 to 428.82]
  6M PVT-Slo10%RT Moderate OSA | 406.17 [383.96 to 429.66] | 406.78 [385.63 to 429.09]
  6M PVT-Slo10%RT Severe OSA | 394.48 [377.66 to 412.05] | 405.04 [384.90 to 426.24]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M A/P Function- PVT-Slo10%RT. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ. Months since randomization were also included as covariate; Test type: Superiority or Other; p = 0.9656, Mixed Models Analysis — 2M A/P Function- PVT-Slo10%RT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.6765, Mixed Models Analysis — 2M A/P Function- PVT-Slo10%RT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.5288, Mixed Models Analysis — 2M A/P Function- PVT-Slo10%RT (Severe OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.7807, Mixed Models Analysis — 6M A/P Function- PVT-Slo10%RT (Mild OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.9603, Mixed Models Analysis — 6M A/P Function- PVT-Slo10%RT (Moderate OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3075, Mixed Models Analysis — 6M A/P Function- PVT-Slo10%RT (Severe OSA); P<0.05 indicates statistical significance for P values. Data were reciprocal transformed for analysis and back-transformed for reporting; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)

7. Secondary Outcome: Learning and Memory (L/M) Function: Buschke Selective Reminding Test Delayed Recall- Total Recall (BSRTDR-TotRec)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. One of the selected variables came from the domain of Learning and Memory (L/M) Function: Buschke Selective Reminding Test Delayed Recall- Total Recall (BSRTDR-TotRec).
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: number of words recalled
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
number of words recalled
  2M BSRTDR-TotRec Mild OSA | 8.54 [7.99 to 9.10] | 8.20 [7.53 to 8.87]
  2M BSRTDR-TotRec Moderate OSA | 8.49 [8.13 to 8.85] | 8.22 [7.82 to 8.62]
  2M BSRTDR-TotRec Severe OSA | 8.48 [8.20 to 8.76] | 8.21 [7.92 to 8.51]
  6M BSRTDR-TotRec Mild OSA | 9.01 [8.47 to 9.54] | 9.44 [8.92 to 9.97]
  6M BSRTDR-TotRec Moderate OSA | 8.56 [8.14 to 8.98] | 8.91 [8.54 to 9.28]
  6M BSRTDR-TotRec Severe OSA | 8.87 [8.58 to 9.16] | 8.75 [8.48 to 9.01]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M L/M Function- BSRTDR-TotRec. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ. A pre-randomization baseline BSRTDR-TotRec was also included as a covariate; Test type: Superiority or Other; p = 0.4262, Regression, Linear — 2M L/M Function- BSRTDR-TotRec (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3161, Regression, Linear — 2M L/M Function- BSRTDR-TotRec (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1835, Regression, Linear — 2M L/M Function- BSRTDR-TotRec (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.2462, Regression, Linear — 6M L/M Function- BSRTDR-TotRec (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.2069, Regression, Linear — 6M L/M Function- BSRTDR-TotRec (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5235, Regression, Linear — 6M L/M Function- BSRTDR-TotRec (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)

8. Secondary Outcome: Executive and Frontal-Lobe (E/F) Function: Sustained Working Memory Test- Mid-day Behavioral Index (SWMT-BehMD)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Executive and Frontal-Lobe (E/F) Function: SWMT-BehMD, SWMT-ActMD, and SAT-D-NumRuCh.
  These data are for variable #1: Sustained Working Memory Test- Mid-day Behavioral Index (SWMT-BehMD)
  SWMT-BehMD is a scaled score that indicates whether the participant scored lower or higher relative to baseline using standard deviation units. It is computed as the difference from baseline relative to measures of working memory (WM) task performance accuracy (percent correct) and mean and standard deviation of reaction time (milliseconds). High-load WM tasks receive twice the weight of the low-load WM tasks.
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
score on a scale
  2M SWMT-BehMD Mild OSA | 0.180 [0.006 to 0.355] | 0.104 [-0.074 to 0.283]
  2M SWMT-BehMD Moderate OSA | 0.137 [0.035 to 0.238] | 0.126 [0.007 to 0.245]
  2M SWMT-BehMD Severe OSA | 0.205 [0.117 to 0.294] | -0.011 [-0.128 to 0.106]
  6M SWMT-BehMD Mild | 0.143 [-0.072 to 0.357] | 0.116 [-0.123 to 0.356]
  6M SWMT-BehMD Moderate OSA | 0.194 [0.062 to 0.325] | 0.314 [0.191 to 0.437]
  6M SWMT-BehMD Severe OSA | 0.321 [0.212 to 0.430] | 0.173 [0.052 to 0.295]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M E/F Function- SWMT-BehMD. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ; Test type: Superiority or Other; p = 0.5419, Regression, Linear — 2M E/F Function- SWMT-BehMD (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.8900, Regression, Linear — 2M E/F Function- SWMT-BehMD (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0031, Regression, Linear — 2M E/F Function- SWMT-BehMD (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 6M E/F Function- SWMT-BehMD. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ; Test type: Superiority or Other; p = 0.8703, Regression, Linear — 6M E/F Function- SWMT-BehMD (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.1838, Regression, Linear — 6M E/F Function- SWMT-BehMD (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.0739, Regression, Linear — 6M E/F Function- SWMT-BehMD (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)

9. Secondary Outcome: Executive and Frontal-Lobe (E/F) Function: SWMT- Mid-day Activation Index (SWMT-ActMD)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Executive and Frontal-Lobe (E/F) Function: SWMT-BehMD, SWMT-ActMD, and SAT-D-NumRuCh.
  These data are for variable #2: SWMT- Mid-day Activation Index (SWMT-ActMD)
  SWMT-ActMD is a scaled score that indicates whether the participant scored lower or higher relative to baseline (BL) using standard deviation units. It is computed as the difference from BL relative to EEG power spectral variables (decibels) measured during the easier vs. more difficult working memory (WM) tasks. A positive activation sub-score indicates a larger cortical neuronal population was recruited to perform the more difficult WM task relative to BL, while a negative score indicates a smaller population was recruited.
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
score on a scale
  2M SWMT-ActMD Mild | -0.050 [-0.268 to 0.169] | 0.317 [0.031 to 0.603]
  2M SWMT-ActMD Moderate OSA | 0.262 [0.084 to 0.440] | 0.170 [0.006 to 0.334]
  2M SWMT-ActMD Severe OSA | -0.003 [-0.109 to 0.103] | 0.033 [-0.093 to 0.159]
  6M SWMT-ActMD Mild | 0.157 [-0.089 to 0.403] | 0.118 [-0.117 to 0.353]
  6M SWMT-ActMD Moderate OSA | 0.016 [-0.131 to 0.162] | 0.014 [-0.188 to 0.216]
  6M SWMT-ActMD Severe OSA | 0.058 [-0.068 to 0.185] | 0.123 [-0.016 to 0.262]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M E/F Function- SWMT-ActMD. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ; Test type: Superiority or Other; p = 0.0450, Regression, Linear — 2M E/F Function- SWMT-ActMD (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.4512, Regression, Linear — 2M E/F Function- SWMT-ActMD (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.6672, Regression, Linear — 2M E/F Function- SWMT-ActMD (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 6M E/F Function- SWMT-ActMD. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ; Test type: Superiority or Other; p = 0.8197, Regression, Linear — 6M E/F Function- SWMT-ActMD (Mild OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.9890, Regression, Linear — 6M E/F Function- SWMT-ActMD (Moderate OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.5029, Regression, Linear — 6M E/F Function- SWMT-ActMD (Severe OSA); P<0.05 indicates statistical significance for P values; Generalized Linear Models (GLM) were run by visit (2M and 6M)

10. Secondary Outcome: Executive and Frontal-Lobe (E/F) Function: Shifting Attention Test Discovery Condition- Number of Rule Changes (SAT-D-NumRuCh)
Description: The APPLES a priori Secondary Neurocognitive Analysis Plan specified a dimension reduction method to reduce twelve secondary neurocognitive variables from three neurocognitive domains to seven variables from three neurocognitive domains. Three of the selected variables came from the domain of Executive and Frontal-Lobe (E/F) Function: Sustained Working Memory Test- Mid-day Behavioral Index (SWMT-BehMD), SWMT- Mid-day Activation Index (SWMT-ActMD), and Shifting Attention Test Discovery Condition- Number of Rule Changes (SAT-D-NumRuCh).
  These data are for variable #3: Shifting Attention Test Discovery Condition- Number of Rule Changes (SAT-D-NumRuCh)
Time Frame: 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: number of rule changes (dichotomized)
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
number of rule changes (dichotomized)
  2M SAT-D-NumRuCh Mild OSA | 0.931 [0.885 to 0.977] | 0.929 [0.873 to 0.985]
  2M SAT-D-NumRuCh Moderate OSA | 0.936 [0.904 to 0.968] | 0.951 [0.924 to 0.979]
  2M SAT-D-NumRuCh Severe OSA | 0.952 [0.931 to 0.972] | 0.942 [0.918 to 0.967]
  6M SAT-D-NumRuCh Mild | 0.897 [0.827 to 0.966] | 0.907 [0.832 to 0.982]
  6M SAT-D-NumRuCh Moderate OSA | 0.903 [0.853 to 0.953] | 0.935 [0.896 to 0.975]
  6M SAT-D-NumRuCh Severe OSA | 0.927 [0.894 to 0.959] | 0.924 [0.888 to 0.960]
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for covariate adjusted 2M E/F Function- SAT-D-NumRuCh. Covariates were designated in the a priori secondary analysis plan as being the most likely to explain variation in the outcomes. Covariates included: study arm, OSA severity, sex, race, % of total sleep time oxygen saturation < 85% (PSG), age < 60 years, WASI Verbal IQ, and WASI Performance IQ; Test type: Superiority or Other; p = 0.9518, Mixed Models Analysis — 2M E/F Function- SAT-D-NumRuCh (Mild OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.4108, Mixed Models Analysis — 2M E/F Function- SAT-D-NumRuCh (Moderate OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.4528, Mixed Models Analysis — 2M E/F Function- SAT-D-NumRuCh (Severe OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.8391, Mixed Models Analysis — 6M E/F Function- SAT-D-NumRuCh (Mild OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.2771, Mixed Models Analysis — 6M E/F Function- SAT-D-NumRuCh (Moderate OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.8961, Mixed Models Analysis — 6M E/F Function- SAT-D-NumRuCh (Severe OSA); P<0.05 indicates statistical significance for P values. Outcome formulated as dichotomized variable (<=2 vs. >=3) based on a 5th percentile cut-off used in pilot studies per test developer suggestion; Generalized Linear Mixed Models (GLMM) were utilized to account for repeated measures (DX, 2M, 6M)

11. Secondary Outcome: Objective Sleepiness/Alertness: Maintenance of Wakefulness Test- Mean Sleep Latency (MWT-MSL)
Description: Objective sleepiness/alertness was measured using the Maintenance of Wakefulness Test (MWT); the outcome variable was MWT Mean Sleep Latency (MWT-MSL).
  The MWT was administered using four twenty-minute trials where the participant was asked to sit in a chair, in a quiet and dimly lit room, with instructions to stay awake. Trials were performed at 10 AM, Noon, 2 PM and 4 PM. The mean sleep latency was calculated using the 4 trials from a given visit, and required that at least 3 of the 4 trials were performed and validated.
Time Frame: Measured at diagnostic visit (baseline) and 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
minutes
  DX MWT-MSL | 17.13 (3.86) | 16.95 (4.13)
  DX MWT-MSL Mild OSA | 17.51 (3.71) | 17.62 (3.38)
  DX MWT-MSL Moderate OSA | 17.74 (3.50) | 17.76 (3.68)
  DX MWT-MSL Severe OSA | 16.68 (4.05) | 16.35 (4.43)
  2M MWT-MSL | 17.96 (3.40) | 17.27 (3.89)
  2M MWT-MSL Mild OSA | 17.52 (3.60) | 18.21 (2.94)
  2M MWT-MSL Moderate OSA | 17.91 (3.39) | 18.14 (2.93)
  2M MWT-MSL Severe OSA | 18.10 (3.35) | 16.63 (4.34)
  6M MWT-MSL | 18.11 (3.27) | 17.34 (3.82)
  6M MWT-MSL Mild OSA | 17.77 (4.00) | 17.89 (3.27)
  6M MWT-MSL Moderate OSA | 17.90 (3.41) | 18.18 (3.27)
  6M MWT-MSL Severe OSA | 18.30 (2.98) | 16.78 (4.10)
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.6540, Chop-lump Wilcoxon — DX- MWT-MSL; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.9778, Chop-lump Wilcoxon — DX- MWT-MSL (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.8314, Chop-lump Wilcoxon — DX- MWT-MSL (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.5018, Chop-lump Wilcoxon — DX- MWT-MSL (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.0052, Chop-lump Wilcoxon — 2M- MWT-MSL; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.2476, Chop-lump Wilcoxon — 2M- MWT-MSL (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 7: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.7520, Chop-lump Wilcoxon — 2M- MWT-MSL (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 8: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.0002, Chop-lump Wilcoxon — 2M- MWT-MSL (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 9: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.0022, Chop-lump Wilcoxon — 6M- MWT-MSL; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 10: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.7630, Chop-lump Wilcoxon — 6M- MWT-MSL (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 11: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.5170, Chop-lump Wilcoxon — 6M- MWT-MSL (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling
Statistical Analysis 12: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Objective Sleepiness/Alertness- MWT-MSL; Test type: Superiority or Other; p = 0.0002, Chop-lump Wilcoxon — 6M- MWT-MSL (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Chop-lump test was selected due to a high frequency of scores at the twenty-minute ceiling

12. Secondary Outcome: Subjective Sleepiness/Alertness: Epworth Sleepiness Scale- Total Score (ESS-TS)
Description: Subjective sleepiness/alertness was measured using the Epworth Sleepiness Scale (ESS); the outcome variable was ESS Total Score (ESS-TS).
  The ESS is a validated questionnaire (8 questions) that ask the chances of dozing off in specific situations. Summing the scores produces a scaled total score between 0 and 24, with higher numbers indicating more subjective sleepiness. The ESS was administered the evening before the polysomnogram (PSG), or overnight sleep study. Data reported here include questionnaires collected at the DX, 2M, and 6M visits.
Time Frame: Measured at diagnostic visit (baseline) and 2 months and 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 556 | 542
scores on a scale
  DX ESS-TS | 10.07 (4.26) | 10.09 (4.39)
  DX ESS-TS Mild OSA | 10.10 (4.55) | 9.73 (4.43)
  DX ESS-TS Moderate OSA | 9.57 (4.13) | 9.75 (4.56)
  DX ESS-TS Severe OSA | 10.35 (4.24) | 10.37 (4.28)
  2M ESS-TS | 7.86 (4.20) | 8.89 (4.31)
  2M ESS-TS Mild OSA | 8.59 (4.31) | 7.90 (4.01)
  2M ESS-TS Moderate OSA | 7.25 (3.89) | 8.39 (4.29)
  2M ESS-TS Severe OSA | 8.00 (4.31) | 9.34 (4.34)
  6M ESS-TS | 7.39 (4.21) | 8.41 (4.18)
  6M ESS-TS Mild OSA | 8.37 (4.64) | 7.64 (3.98)
  6M ESS-TS Moderate OSA | 7.07 (3.87) | 8.43 (4.55)
  6M ESS-TS Severe OSA | 7.31 (4.25) | 8.56 (4.02)
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.9291, Regression, Linear — DX- ESS-TS; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 2: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.6152, Regression, Linear — DX- ESS-TS (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 3: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.7040, Regression, Linear — DX- ESS-TS (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 4: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for DX Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.9537, Regression, Linear — DX- ESS-TS (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 5: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0004, Regression, Linear — 2M- ESS-TS; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 6: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.3886, Regression, Linear — 2M- ESS-TS (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 7: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0236, Regression, Linear — 2M- ESS-TS (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 8: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 2M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0005, Regression, Linear — 2M- ESS-TS (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 9: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0005, Regression, Linear — 6M- ESS-TS; Comparison of means by visit only; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 10: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.3796, Regression, Linear — 6M- ESS-TS (Mild OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 11: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0106, Regression, Linear — 6M- ESS-TS (Moderate OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution
Statistical Analysis 12: Comparison: Active CPAP vs Sham CPAP; Comparison of means (regression estimates) between arms for 6M Subjective Sleepiness/Alertness- ESS-TS; Test type: Superiority or Other; p = 0.0010, Regression, Linear — 6M- ESS-TS (Severe OSA); Comparison of means by visit and Obstructive Sleep Apnea (OSA) severity; P<0.05 indicates statistical significance for P values; Regression analyses for the ESS used Generalized Linear Models (GLM) for an over-dispersed binomial distribution

13. Secondary Outcome: Mood
Time Frame: Measured at diagnostic visit (baseline) and 2 months and 6 months post intervention
Population: Mood was dropped as a secondary outcome measure for analysis by our Core Team.
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Quality of Life: Calgary Sleep Apnea Quality of Life Index- Total Score (SAQLI-TS)
Description: Quality of life was measured using the Calgary Sleep Apnea Quality of Life Index (SAQLI), which is an interview-administered instrument with high internal consistency and reliability. The SAQLI was designed to assess components identified as important to patients including daily functioning, social interactions, emotional functioning, symptoms experienced, and treatment-related symptoms. Items are scored on a seven-point scale, averaged (taking into account treatment-related symptoms), to yield a composite score between 1 and 7, where higher scores represent better quality of life.
Time Frame: diagnostic visit (baseline)
Population: Analyses performed for group of participants with SAQLI data. Baseline demographics were generally similar (mean age, sex ratio, proportion of white participants, average body mass index), and participants in both groups had similar SAQLI scores at baseline, which are presented below.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 443 | 402
Units on a scale | 4.7 (0.8) | 4.7 (0.8)

15. Other Pre Specified Outcome: Functional Magnetic Resonance Imaging (fMRI)
Time Frame: Measured at diagnostic visit (baseline) and 6 months post intervention
Population: fMRI was dropped as a secondary outcome measure for analysis by our Core Team.
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from participant enrollment though the end of study visit (6 months). The APPLES Data and Safety Monitoring Board (DSMB) indicated events should be reported by body systems/event categories; data are reported this way.
Description: All Serious Adverse Events (SAEs) and Adverse Events (AEs) were categorized into 17 body systems/event categories. Safety data were reviewed regularly by the APPLES DSMB; three categories were deemed most important for SAEs: Cardiovascular, MVA, and Death. Analyses were performed on post-randomization events.
Arm/Group | Active CPAP | Sham CPAP
Serious Adverse Events (participants affected / at risk) | 32/556 | 31/542
Other Adverse Events (participants affected / at risk) | 390/556 | 373/542
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=556) | Sham CPAP (N=542)
Cardiovascular (Cardiac disorders) | 4 (4) | 6 (7)
Motor Vehicle Accident (MVA) (General disorders) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
General (General disorders) | 2 (2) | 3 (3)
Genitourinary (Renal and urinary disorders) | 0 (0) | 4 (4)
GI / Digestive (Gastrointestinal disorders) | 6 (6) | 5 (5) — Gastrointestinal / Digestive
HEENT (General disorders) | 1 (1) | 1 (1) — Head, eyes, ears, nose, and throat
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 13 (13) | 5 (5)
Near-miss MVA (General disorders) | 0 (0) | 3 (3) — Near-miss Motor Vehicle Accident
Neurological (Nervous system disorders) | 3 (3) | 0 (0)
Other accident (General disorders) | 1 (1) | 3 (3)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=556) | Sham CPAP (N=542)
Cardiovascular (Cardiac disorders) | 27 (29) | 23 (28)
Motor Vehicle Accident (MVA) (General disorders) | 10 (10) | 11 (11)
Dermatological (Skin and subcutaneous tissue disorders) | 101 (125) | 61 (75)
Endocrinological (Endocrine disorders) | 7 (7) | 3 (3)
General (General disorders) | 52 (58) | 36 (42)
Genitourinary (Renal and urinary disorders) | 13 (13) | 14 (14)
GI / Digestive (Gastrointestinal disorders) | 32 (36) | 28 (30) — Gastrointestinal / Digestive
HEENT (General disorders) | 207 (269) | 154 (191) — Head, eyes, ears, nose, and throat
Hematologic / Lymphatic (Immune system disorders) | 3 (3) | 3 (5)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 44 (61) | 45 (53)
Near-miss MVA (General disorders) | 7 (7) | 8 (8) — Near-miss Motor Vehicle Accident
Neurological (Nervous system disorders) | 33 (36) | 32 (36)
Psychiatric (Psychiatric disorders) | 42 (48) | 59 (69)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 135 (186) | 153 (185)
Other Accident (General disorders) | 20 (21) | 25 (25)
Work-related Accident (General disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
There are study sample limitations because although participants with severe OSA were included, those who had the lowest oxygen saturation, a history of sleepiness-related accidents, or major cardiovascular comorbidities were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No